CLINICAL TRIAL: NCT02293408
Title: A Prospective Cross-Sectional and Longitudinal Study With Additional Retrospective Chart Review to Evaluate Clinical and Biochemical Characteristics and Disease Progression in Patients With Mucopolysaccharidosis Type IIIB
Brief Title: Natural History Study to Characterise the Course of Disease Progression in Participants With Mucopolysaccharidosis Type IIIB
Status: Terminated | Type: Observational
Why Stopped: The Sponsor's decision to terminate the SBC-103 program was reached after review of the data from all interventional clinical studies of SBC-103.
Sponsor: Alexion Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: NGLU-NH02
Record Dates: First submitted 2014-11-03; First posted 2014-11-18 (Estimated); Last update posted 2018-09-13 (Actual); Status verified 2018-09

CONDITIONS: MPS IIIB (Sanfilippo B Syndrome)
Keywords: MPS IIIB; Mucopolysaccharidosis; Mucopolysaccharidosis type IIIB; Sanfilippo Syndrome Type B
MeSH Terms: conditions — Mucopolysaccharidosis III; Mucopolysaccharidoses

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Clinical laboratory tests, including heparan sulfate and exploratory disease biomarkers from serum and urine.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Component 1: Component 1 involved an evaluation of the clinical characteristics of MPS IIIB in participants based on a retrospective chart review to collect information on demographics, clinical history, diagnostic tests, treatments, clinical chemistry and hematology test results, physical examination findings, anthropometric data, radiology results, and supportive interventions performed over a period of up to 6 weeks.
- Component 2: Component 2 involved a longitudinal evaluation of the course of disease progression in a subset of participants considered to be at risk of rapid disease progression, who, after completing Component 1, were to be prospectively followed for a period of at least 1 year (Longitudinal Follow-Up) and up to 3 years total (Extended Follow-Up).

SUMMARY:
The objectives of this study are to describe the clinical and biochemical characteristics and course of disease progression in participants with Mucopolysaccharidosis type IIIB (MPS IIIB)

ELIGIBILITY:
Inclusion Criteria:

A participant must meet all of the following inclusion criteria to be eligible for this study:

1. The participant has a definitive diagnosis of MPS IIIB, as determined by either of the following:

   1. Documented deficiency in alpha-N-acetyl-glucosaminidase (NAGLU) enzyme activity or
   2. Documented functionally-relevant mutations in both alleles of the NAGLU gene.
2. The participant is at least 1 year of age (biological age).
3. The participant or the participant's parent provides informed consent.
4. The participant is willing and able to comply with protocol requirements to the extent that may be expected of a participant with cognitive impairment.

In addition to the eligibility criteria above, a participant must meet all of the following criteria for Component 2:

1. The participant meets criterion a or criterion b below.

   a. The participant is considered to be at risk of rapid disease progression based on at least 1 of the following criteria:

   i. The participant has documented mutations of the NAGLU gene that are reported to be linked to rapid disease progression (for example, disease onset before 6 years of age), or

   ii. The participant has a sibling, or other first- or second-degree relative with rapidly progressing MPS IIIB (for example, disease onset before 6 years of age).

   b. The participant had disease onset prior to 6 years of age (biological age), as defined by:

   i. Cognitive delay evaluated by Bayley Scales of Infant Development, Third Edition (BSID-III) or Kaufman Assessment Battery for Children, Second Edition (KABC-II), or

   ii. Language delay, plateauing, or regression of language skills as determined by the Investigator (for example, participant uses isolated words, associated words such as 2-word combinations, sentences, poor or reduced language, and/or difficult to understand).
2. The participant has an age equivalent of ≥1 year on the Vineland Adaptive Behavior Scales, Second Edition (Vineland II).

Exclusion Criteria:

A participant who meets any of the following exclusion criteria will be ineligible for this study:

1. The participant has visual or hearing impairments sufficient to preclude cooperation with neurodevelopmental testing.
2. The participant has a history of poorly-controlled seizure disorder.
3. The participant is currently receiving medication, which, in the Investigator's opinion, would be likely to substantially confound interpretation of the results (for example, the participant has been on the current dose of psychotropic medication for less than 3 months).
4. The participant is receiving a newly increased dose of melatonin (for example, less than 3 months on current dose).
5. The participant has previously received an investigational therapy for MPS IIIB (with the exception of high dose Genistein >150 milligram/kilogram (mg/kg)/day, which will require a minimum of 3 months wash-out before entering the study) or has had hematopoietic stem cell transplant (HSCT).
6. The participant has any other prior or ongoing medical condition that may present a safety risk, interfere with study compliance, or confound data interpretation.

Min Age: 1 Year | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: 27 participants with MPS IIIB were enrolled and analyzed in Component 1.
  Component 1 (27 participants): The participant has a definitive diagnosis of MPS IIIB. Component 2 (15 participants from Component 1): The participant is considered to be at risk of rapid disease progression.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2014-09-14 (Actual); Primary Completion 2017-07-11 (Actual); Study Completion 2017-07-11 (Actual)

PRIMARY OUTCOMES:
Collection And Analysis Of Clinical Characteristics Of MPS IIIB | Baseline to Week 43
  Component 1 involved an evaluation of the clinical characteristics of MPS IIIB in participants based on a retrospective chart review to collect information on demographics, clinical history, diagnostic tests, treatments, clinical chemistry and hematology test results, physical examination findings, anthropometric data, radiology results, and supportive interventions performed over a period of up to 6 weeks.
Longitudinal Analysis Of The Course Of Disease Progression In Participants With MPS IIIB | Baseline to Week 43
  Component 2 involved a longitudinal evaluation of the course of disease progression in a subset of participants considered to be at risk of rapid disease progression, who, after completing Component 1, were to be prospectively followed for a period of at least 1 year (Longitudinal Follow-Up) and up to 3 years total (Extended Follow-Up).

CONTACTS AND LOCATIONS:
Locations (7):
- United States (2):
  - Minneapolis, Minnesota
  - Pittsburgh, Pennsylvania
- Porto Alegre, Brazil
- Monza, Italy
- Coimbra, Portugal
- Barcelona, Spain
- Birmingham, United Kingdom